CLINICAL TRIAL: NCT01500447
Title: The Molecular Basis of Inherited Reproductive Disorders
Brief Title: Inherited Reproductive Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120049; 12-E-0049
Record Dates: First submitted 2011-12-21; First posted 2011-12-28 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Genetic Disorder; Infertility; Hypogonadism; Amenorrhea
Keywords: Hypogonadotropic Hypogonadism; Kallmann Syndrome; Delayed Puberty; Hypothalamic Amenorrhea; Precocious Puberty; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn; Infertility; Hypogonadism; Amenorrhea; Kallmann Syndrome; Puberty, Delayed; Puberty, Precocious

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central Precious Puberty: CPP subjects
- Hypogonadotropic Hypogonadism: IHH, KS, GnRH Deficiency, BAM syndrome (arhinia), HA, CDP subjects

SUMMARY:
Background:

- During puberty, children begin to develop into adults. Problems with the hormones released during puberty can affect the reproductive system. Some people have low hormone levels that severely delay or prevent puberty. Others start puberty abnormally early. Other people may have a normal puberty but develop reproductive disorders later in life. Researchers want to study people with reproductive disorders to learn more about how these disorders may be inherited.

Objectives:

- To learn how reproductive system disorders may be inherited.

Eligibility:

* People with one of the following problems:
* Abnormally early puberty
* Abnormally late or no puberty
* Normal puberty with hormonal problems that develop later in life
* People who have not yet had puberty but have symptoms that indicate low hormone levels.

Design:

* Participants will provide a blood sample for testing. They will complete a questionnaire about their symptoms. They will also have a scratch-and-sniff test to study any problems with their ability to smell.
* Participant medical records will be reviewed. Participants will also provide a family medical history.
* Family members of those in the study may be invited to participate.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
The key initiating factors for reproductive development remain among the great mysteries of pediatric and reproductive endocrinology. The onset of puberty is initiated by pulsatile secretion of gonadotropin-releasing hormone (GnRH) from the hypothalamus. The neuroendocrine events leading to increased GnRH secretion and the resultant onset of puberty remain largely unknown.

Isolated deficiency of GnRH results in the rare clinical syndrome of idiopathic hypogonadotropic hypogonadism (IHH), where decreased secretion of GnRH results in impaired gonadotropin secretion. The resultant hypogonadism presents with delayed, incomplete, or absent sexual maturation. Human and animal models have identified a number of genes responsible for IHH, but more than half of patients with clinical evidence of the disorder do not have a detectable mutation. In addition, there is significant clinical heterogeneity among affected individuals, including members of the same family harboring the same mutations. Careful human phenotyping of such patients and families has expanded our understanding of this spectrum of disorders to include oligo-digenic inheritance, as well as reversibility of the condition, and has provided insight into developmental pathways involved in the ontogeny of GnRH neurons. In particular, hypogonadotropic hypogonadism (HH) exists along a genetic and phenotypic spectrum that includes milder forms of GnRH dysregulation, precocious and delayed puberty, and onset of reproductive dysfunction after puberty.

Genetic analysis of subjects with unknown mutations is likely to yield important insights into additional pathways involved in the regulation of GnRH secretion. Here, we propose a genetic investigation of subjects with IHH to characterize further the phenotypic effects of previously described genetic variants, as well as to identify novel genes involved in congenital GnRH deficiency. We will use candidate gene and whole exome approaches, as well as linkage analysis.

This protocol will utilize the disease model of IHH to increase our understanding of the physiology of GnRH secretion, including the neuroendocrine regulation of GnRH pulsatility. Examining the genetic characteristics of subjects with isolated GnRH deficiency will reveal insights into the mechanisms underlying the reawakening of the hypothalamic-pituitary-gonadal axis at puberty, providing opportunities for new diagnostic capabilities and therapeutic interventions for disorders of puberty and fertility.

ELIGIBILITY:
* INCLUSION CRITERIA:

The essential inclusion criteria include:

1. failure to go through a normal, age-appropriate, spontaneous puberty and low sex steroid levels in the setting of low/normal gonadotropins (due to substantial variability among patient presentations, this will be based on the clinical judgement of the Investigator), or
2. abnormally early development of puberty, or
3. normal puberty with subsequent development of low gonadotropin levels, or
4. individuals with features indicating an increased risk of hypogonadotropic hypogonadism.
5. Family members: both affected and unaffected family members are strongly encouraged to participate.

EXCLUSION CRITERIA:

Since hypogonadotropic hypogonadism is a rare condition, this protocol remains open to enrollment so that we may study all subjects that are both qualified and interested in participating.

Because HH represents a spectrum, where associated clinical findings may provide phenotypic clues to the assessment of inheritability and underlying physiology, exclusion criteria are very limited:

* Patients who have additional pituitary deficiencies, effectively ruling out isolated GnRH deficiency, whether these deficiencies are congenital or acquired (e.g. secondary to malignancy, infection, or irradiation).
* Patients who are taking medications known to affect GnRH secretion, such as corticosteroids or continuous opiate administration (or were taking them at the time of diagnosis).

Ages: 6 Weeks to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Clinical, self-referred or physician-referred subjects
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2012-04-25 (Actual)

PRIMARY OUTCOMES:
The main outcome is the identification of known and novel genetic variants in individuals representing the complete spectrum of idiopathic hypogonadotropic hypogonadism. | Ongoing/exploratory
  The main outcome is the identification of known and novel genetic variants in individuals representing the complete spectrum of idiopathic hypogonadotropic hypogonadism.

SECONDARY OUTCOMES:
Phenotypic correlations, made by comparing the results of the genotypic analysis with clinical and/or biochemical characteristics, as well as the discovery of genes worthy of further functional analysis. | Ongoing/exploratory
  Phenotypic correlations, made by comparing the results of the genotypic analysis with clinical and/or biochemical characteristics, as well as the discovery of genes worthy of further functional analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D Shaw, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
This study does not meet the criteria of a clinical trial, therefore ICMJE does not require a data sharing statement.@@@@@@@@@@@@The study will comply with the NIH Genomic Data Sharing Policy, if in the future, it meets the Policy s criteria for large scale human genomic data.

REFERENCES:
- [Derived] Delaney A, Burkholder AB, Lavender CA, Plummer L, Mericq V, Merino PM, Quinton R, Lewis KL, Meader BN, Albano A, Shaw ND, Welt CK, Martin KA, Seminara SB, Biesecker LG, Bailey-Wilson JE, Hall JE. Increased Burden of Rare Sequence Variants in GnRH-Associated Genes in Women With Hypothalamic Amenorrhea. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1441-e1452. doi: 10.1210/clinem/dgaa609. PMID 32870266
- [Derived] Meader BN, Albano A, Sekizkardes H, Delaney A. Heterozygous Deletions in MKRN3 Cause Central Precocious Puberty Without Prader-Willi Syndrome. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2732-9. doi: 10.1210/clinem/dgaa331. PMID 32480405
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-E-0049.html